CLINICAL TRIAL: NCT06107920
Title: Neoadjuvant Chemotherapy for Obstructive Colon cancER First Treated by cOlostomy : A Randomized Phase III Trial - COnCERTO (French 01-18)
Brief Title: Neoadjuvant Chemotherapy for Obstructive Colon cancER First Treated by cOlostomy
Acronym: COnCERTO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/0407/HP
Record Dates: First submitted 2023-10-25; First posted 2023-10-30 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Adjuvant chemotherapy) / Control arm (No Intervention): Diverting stoma - colectomy - +/- adjuvant chemotherapy
  The colectomy (open or laparoscopic) should be performed within 1 to 20 days after the randomization and with respect of the oncological quality criteria of resection. After completion of surgery, adjuvant chemotherapy will be discussed as follow:
  * Low-risk stage II: No adjuvant treatment
  * High-risk MSS stage II (vascular emboli, lymphatic or perinervous invasion, poor differentiation, <12 harvested lymph nodes, perforation): Investigator's discretion
  * pT1-T3N1: CAPOX (3 months) or FOLFOX (6 months)
  * pT4 and/or N2: FOLFOX (6 months)
- Arm II (Neoadjuvant Chemotherapy) / Experimental arm (Experimental): Patients receive systemic CAPOX or FOLFOX chemotherapy (3 months) within 21 days after the randomization. After completion of neoadjuvant chemotherapy and within 3 to 5 weeks, the colectomy (open or laparoscopic) will be performed with respect of the oncological quality criteria. Adjuvant chemotherapy will be discussed as follow:
  * Low-risk stage II: No adjuvant treatment
  * High-risk MSS stage II (vascular emboli, perinervous or lymphatic invasion, poor differentiation, <12 harvested lymph nodes, perforation): Investigator's discretion
  * Stage III: CAPOX or FOLFOX (3 months)
  Interventions: Drug: Neoadjuvant chemotherapy

INTERVENTIONS:
Drug: Neoadjuvant chemotherapy — Diverting stoma- neoadjuvant chemotherapy - colectomy - +/- adjuvant chemotherapy
  Other Names: Arm II
  Arms: Arm II (Neoadjuvant Chemotherapy) / Experimental arm

SUMMARY:
The aim of this study is to determine whether chemotherapy prior to tumor removal (neoadjuvant chemotherapy), in patients undergoing treatment for colon cancer in occlusion (CCO), would improve the rate of patients able to benefit from "optimal" treatment, i.e. complete treatment (including all neoadjuvant and adjuvant chemotherapy cures).

This new strategy, which would combine chemotherapy before surgery and possibly post-operatively (depending on tumor analysis), could improve the prognosis of occluded colon cancers by treating circulating micrometastases and/or inducing a reduction in tumor size, thereby increasing the rate of complete resection.

DETAILED DESCRIPTION:
In France, for patients admitted for an obstructive colon cancer, surgery is the preferred strategy. Primary diverting stoma is associated with low morbidity, and low 30-day mortality. Primary diverting stoma is not a major surgical undertaken, is effective to relief bowel obstruction, enables optimization of the patient's condition, allows adequate oncological staging and secondary elective colectomy. This strategy is actually recommended by the French and European Guidelines in patients with left-sided obstructive colon cancer and may be an option in patients with right-sided obstructive colon cancer, especially in those at high risk of postoperative complications

Urgent surgery for obstructive colon cancer is associated with increased risk of postoperative morbidity, mortality and permanent stoma rates as it is generally performed in elderly patients with poor medical condition or in patients with severe comorbidities. Moreover, obstructive colon cancers are diagnosed at locally advanced (T4) or metastatic stage and, at equal tumour stage, obstruction itself negatively impacts oncological outcomes in colon cancer patients. Among the several factors that may explain poor oncological outcomes of OCC, the absence of adjuvant chemotherapy may play an important role.

Adjuvant chemotherapy is the standard of care for patients undergoing curative resection for a stage III CC. For those with MSS high-risk stage II CC, adjuvant treatment is still a matter of debate. However, in the particular setting of MSS stage II obstructing CC, adjuvant chemotherapy may improve oncological outcomes. Because of high postoperative morbidity and patients' medical conditions, up to 37% of OCC patients for whom adjuvant systemic chemotherapy is considered appropriate do not receive this treatment. It is our hypothesis that the initiation of chemotherapy before resection of the primary tumour in a perioperative setting in patients with non-metastatic OLCC and for whom the obstruction has been relieved by a colostomy may allow to treat a higher proportion of patients with a full curative therapeutic sequence (including resection and chemotherapy if needed).

Randomized phase II-III trials have demonstrated the feasibility (tolerance, postoperative morbidity) and the efficacy (tumor downstaging, tumor downsizing, histological regression, higher R0 resection rate) of neoadjuvant FOLFOX or CAPOX chemotherapy in uncomplicated colon cancer with a trend towards an improvement of DFS. Data of these studies led the French Oncological Authorities to accept neoadjuvant chemotherapy in a perioperative setting as a therapeutic option in patients with locally advanced colon cancer (TNCD 21/01/2019, chapter 3, Cancer du colon non métastatique (p10): "Neo-adjuvant chemotherapy may be considered for locally advanced tumors deemed unresectable or at the limit of resectability (expert opinion)"; "it is possible to perform an upstream stoma before starting chemotherapy ("neo-adjuvant") and then a re-intervention aimed at exeresis (expert opinion). This treatment option should be discussed at the preoperative multidisciplinary consultation meeting if a T4 tumor is suspected during the preoperative workup."

The authors concluded that neoadjuvant chemotherapy using FOLFOX was feasible and might be a treatment option for patients with obstructive colon cancer for whom the obstruction has been relieved by a definctioning stoma. Further large-scale studies are warranted to confirm the present findings. This is exactly what COnCERTO trial aims to determine.

It is our hypothesis that the initiation of neoadjuvant chemotherapy in a perioperative setting in patients with non-metastatic MSS/pMMR Obstructive Colon Cancer (OCC) and for whom the obstruction has been relieved by a stoma may improve the compliance of the treatment and thus may allow to increase the rate of patients receiving the full curative therapeutic sequence according to the guidelines defined as following:

Resection of the primary tumor WITH:

* Low-risk stage II: NO CHEMOTHERAPY
* High-risk stage II: CHEMOTHERAPY AT INVESTIGATOR'S DISCRETION
* Stage III pT1-T3N1: CAPOX (3 months) or FOLFOX (6 months)
* Stage III pT4 and/or N2: FOLFOX (6 months) MSS High-risk stage II are defined as following: No microsatellite instability and presence of vascular emboli, perinervous or lymphatic invasion, poor differentiation, <12 harvested lymph nodes, perforation).

In addition, once OCC are known to have poor prognosis compared to their non-complicated counterparts, neoadjuvant chemotherapy (before resection of the primary) may improve prognosis of these patients by treating circulating micrometastases or by inducing tumor down-staging and thus improving the R0 resection rate.

We thus designed a randomized phase III trial aiming to assess whether FOLFOX or CAPOX neoadjuvant chemotherapy in a perioperative setting may increase the rate of full curative therapeutic sequence in patients with MSS/pMMR OCC first treated by a defunctionning stoma (figure 5).

Demonstrating the positive impact on complicance to the full curative therapic strategy of perioperative chemotherapy in patients with OCC treated by defunctioning stoma, may change medical practices at a national and international level and may lead to a new standard of care. OCC is a major public health issue with no improvement in prognosis during the past decade. By improving the compliance of treatment of patients with OCC, the present study will ensure public health and economic benefits

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ECOG performance status 0 or 1
* Patients with obstructive colon cancer treated by defunctioning stoma
* Pathologically confirmed adenocarcinoma (≥10 cm from the anal verge- left transverse colon) - MSS/pMMR (microsatellites stable primary tumor) status
* Patient requiring colectomy
* Laboratory data including : White blood cell count ≥ 3.109 /L with Neutrophils ≥ 1,5.109 / L, Platelet count ≥ 100.109 / L, Hemoglobin ≥ 9 g/dL (5,6 mmol/L), Total bilirubin ≤ 1,5 x ULN (upper limit of normal), ASAT and ALAT ≤ 2,5 x ULN, Alkaline phosphatase ≤ 1,5 x ULN, Serum creatinine ≤ 1,5 x ULN (performed 10-15 days prior to randomization).
* Non metastatic colon cancer (lung, liver, peritoneal) on thoracic-abdomino-pelvis CT scan
* Absence of synchronous colorectal cancer
* No prior chemotherapy or abdominal or pelvic irradiation
* No history of colorectal cancer
* No serious medical co-morbidity : uncontrolled inflammatory bowel disease, uncontrolled angina, recent [within the past 6 months] myocardial infarction, or another serious medical condition, judged to compromise ability to tolerate chemotherapy and/or surgery
* Women of childbearing potential with effective contraception will be required during chemotherapy treatment and for 6 months after cessation of chemotherapy treatment and a negative blood pregnancy test by beta-HCG at inclusion.
* Women surgically sterile (absence of ovaries and/or uterus)
* Postmenopausal women: confirmation diagnostic (non-medically induced amenorrhea for at least 12 months prior to the inclusion visit)
* For men participating in the study, contraception is required during the trial and for 6 months after stopping chemotherapy treatment.
* Patient able to comply with the study protocol, in the investigator's judgment
* Patient affiliated with, or beneficiary of a social security (national health insurance) category
* Person informed and having signed his consent

Exclusion Criteria:

* Contraindication to colectomy and/or anesthesia
* Rectal cancer located within 10 cm of the anal verge by endoscopy or under the peritoneal reflection at surgery
* Patient having received radiation therapy prior to surgery
* Metastatic spread at baseline assessment (lung, liver, peritoneal)
* History or current evidence on physical examination of central nervous system disease or; Peripheral neuropathy ≥ grade 1
* Contraindication to study neoadjuvant chemotherapy treatments
* Presence of inflammatory bowel disease, HNPCC syndrome or polyposis Clinically relevant coronary artery disease or history of myocardial infarction in the last 6 months, or high risk of uncontrolled arrhythmia
* Uracilemia ≥ 150 ng/ml (suggestive of complete DPD deficiency)
* Medical, geographical, sociological, psychological or legal conditions that would not permit the patient to complete the study or sign informed consent
* Any significant disease, which, in the investigator's opinion, would exclude the patient from the study.
* Patient is a pregnant (positive blood pregnancy test) or breastfeeding (lactating) woman or intending to become pregnant during the study and for at least 6 months after the treatment termination
* Person deprived of liberty by administrative or judicial decision or placed under judicial protection (guardianship or supervision)
* Simultaneous participation in another interventional research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2031-08 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
the success of a full curative therapeutic | 36 months
  The treatment is complete if all the chemotherapy treatments (adjuvant for arm I / neoadjuvant and adjuvant for arm II) is done.

SECONDARY OUTCOMES:
Neoadjuvant chemotherapy Adverse events | 36 months
  Adverse events (grade 3,4 and 5 toxicity) related to neoadjuvant chemotherapy including those related to the primary tumor
adjuvant chemotherapy adverse events | 36 months
  Adverse events (grade 3, 4 and 5 toxicity) related to adjuvant chemotherapy including those related to the primary tumor
Number of cycles administered of neoadjuvant chemotherapy | 36 months
  Number of cycles administered of neoadjuvant chemotherapy
Rate of primary tumour resection | 36 months
  Rate of primary tumour resection
Quality and completeness of the surgical excision | 36 months
  number of lymph nodes examined, completeness of the mesocolon, margins
Overall morbidity according to the Dindo classification | at 90 days postoperatively.
  according to the Dindo classification
Overall mortality | at 3 years and mortality without stoma at 3 years.
  mortality without relapse
Quality of life evaluated using EORTC QLQ-C30 and QLQ-CR29 dedicated to CRC | at J0, week5 (FOLFOX)/week7 (CAPOX), week9 (FOLFOX) and every 6 months a year
  using EORTC QLQ-C30 and QLQ-CR29 dedicated to CRC

CONTACTS AND LOCATIONS:
Locations (27):
- France (27):
  - Chu Amiens, Amiens
  - Chr Beauvais, Beauvais
  - Chru Besancon, Besançon
  - Aphp Avicenne, Bobigny
  - CHU CAEN, Caen
  - Aphp Antoine Beclere, Clamart
  - Chu Colmar, Colmar
  - Chu Dijon, Dijon
  - Chu Grenoble, Grenoble
  - Aphp Kremlin Bicetre, Le Kremlin-Bicêtre
  - Chru Lille, Lille
  - Chu Limoges, Limoges
  - Aphm La Timone, Marseille
  - Aphm Hopital Nord, Marseille
  - Chru Nancy, Nancy
  - Chu Nantes, Nantes
  - Aphp Saint Antoine, Paris
  - Aphp Cochin, Paris
  - Aphp Georges Pompidou, Paris
  - Gh Diaconesses Croix St Simon, Paris
  - CHU LYON, Pierre-Bénite
  - Ch Poissy, Poissy
  - Chu Rouen, Rouen
  - Ch St Denis, Saint-Denis
  - Chu Strasbourg, Strasbourg
  - Chu Tours, Tours
  - Ch Versailles, Versailles

IPD SHARING:
Plan to Share IPD: No